CLINICAL TRIAL: NCT05075421
Title: Comparison of the Prognostic Values of Preoperative Inflammation-based Indices in Patients Undergoing Resection of Gastric Cancer
Brief Title: Prognostic Values of Inflammation-based Indices in Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Suleyman Utku Celik, Principal Investigator, Gulhane Training and Research Hospital
Other Study IDs: Gulhane2021-69
Record Dates: First submitted 2021-10-02; First posted 2021-10-12 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; Survival; Prognosis; Systemic inflammatory response; Markers
MeSH Terms: conditions — Stomach Neoplasms | interventions — Gastrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 (high marker): Patients with elevated serum markers
  Interventions: Procedure: Gastrectomy
- Group 2 (normal marker): Patients with normal value of serum markers
  Interventions: Procedure: Gastrectomy

INTERVENTIONS:
Procedure: Gastrectomy — Any type of gastrectomy for gastric cancer

SUMMARY:
This study aims to evaluate the prognostic values of preoperative inflammation-based indices in patients undergoing potentially curative resection of gastric cancer.

DETAILED DESCRIPTION:
Gastric cancer is one of the most common and deadly cancers worldwide. Based on GLOBOCAN 2018 data, it is the fifth most common malignancy and the third leading cause of cancer deaths, with an estimated 783,000 deaths in 2018. Despite advances in diagnosis and management strategies, outcomes for patients diagnosed with gastric cancer still remain poor and the five-year survival is approximately %20. In addition, there is marked heterogeneity in the duration of survival among patients. Hence, there are increasing research efforts towards the identification of possible predictive clinical, pathological, or biologic factors to determine more accurate patient stratification, which will improve clinical decision-making and possibly contribute to more rational study design and analysis. Systemic inflammation is known to play a crucial role in the pathogenesis, development, and progression of cancer. Preoperative inflammation-based indices, such as the Glasgow prognostic score (GPS), modified Glasgow prognostic score (mGPS), neutrophil-lymphocyte ratio (NLR), platelet lymphocyte ratio (PLR), prognostic index (PI), prognostic nutritional index (PNI), CRP/albumin ratio, systemic inflammation score (SIS), modified systemic inflammation score (mSIS), have been found to have potential prognostic values in various cancer. Previous studies have suggested that several of these scoring systems may have a role in predicting survival in patients with upper gastrointestinal cancer. These scores are all derived from blood tests that are already routinely performed in clinical practice and thus have the potential to offer valuable additional information that may help to guide patient management. This study aims to evaluate the prognostic values of preoperative inflammation-based indices in patients undergoing potentially curative resection of gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 who underwent a surgical procedure for gastric cancer

Exclusion Criteria:

* Patients < 18 years of age
* Patients with no routine blood examination before surgery or incomplete medical records
* Patients followed up less than 3 months
* Patients with additional malignancy
* Patients having tumors that invading adjacent organs
* Patients with adjacent or distant metastasis
* Patients receiving neoadjuvant therapy (chemo- or radiotherapy)
* Patients with previous malignancy history
* Patients with a clinical evidence of infection
* Patients with a history of preoperative use of anti-inflammatory drugs or immunosuppressive treatment
* Patients with a history of chronic inflammatory disease or autoimmune disease
* Patients who underwent emergency surgical resection
* Patients who have undergone R1/R2 resection or those with positive peripheral margins
* Patients with missing data on follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥ 18 years who underwent a surgical procedure for gastric cancer are included in this study
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
5-year survival rates | 5 years
  The primary clinical outcome of interest is 5-year survival rates.

CONTACTS AND LOCATIONS:
Overall Officials: Suleyman U Celik, Principal Investigator — Gulhane Training and Research Hospital
Locations (1):
- Gulhane Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD

REFERENCES:
- [Background] Wen J, Bedford M, Begum R, Mitchell H, Hodson J, Whiting J, Griffiths E. The value of inflammation based prognostic scores in patients undergoing surgical resection for oesophageal and gastric carcinoma. J Surg Oncol. 2018 Jun;117(8):1697-1707. doi: 10.1002/jso.25057. Epub 2018 May 14. PMID 29761518
- [Background] Crumley AB, McMillan DC, McKernan M, McDonald AC, Stuart RC. Evaluation of an inflammation-based prognostic score in patients with inoperable gastro-oesophageal cancer. Br J Cancer. 2006 Mar 13;94(5):637-41. doi: 10.1038/sj.bjc.6602998. PMID 16479253
- [Background] Crumley AB, McMillan DC, McKernan M, Going JJ, Shearer CJ, Stuart RC. An elevated C-reactive protein concentration, prior to surgery, predicts poor cancer-specific survival in patients undergoing resection for gastro-oesophageal cancer. Br J Cancer. 2006 Jun 5;94(11):1568-71. doi: 10.1038/sj.bjc.6603150. PMID 16685271
- [Background] Crumley AB, Stuart RC, McKernan M, Going JJ, Shearer CJ, McMillan DC. Comparison of pre-treatment clinical prognostic factors in patients with gastro-oesophageal cancer and proposal of a new staging system. J Gastrointest Surg. 2010 May;14(5):781-7. doi: 10.1007/s11605-010-1162-6. Epub 2010 Feb 11. PMID 20148314
- [Background] Dutta S, Crumley AB, Fullarton GM, Horgan PG, McMillan DC. Comparison of the prognostic value of tumour and patient related factors in patients undergoing potentially curative resection of gastric cancer. Am J Surg. 2012 Sep;204(3):294-9. doi: 10.1016/j.amjsurg.2011.10.015. Epub 2012 Mar 22. PMID 22444831